CLINICAL TRIAL: NCT04483089
Title: An Observational Real-world Study Evaluating Severe Tricuspid Regurgitation Patients Treated with the Abbott TriClip™ Device
Brief Title: An Observational Real-world Study Evaluating Severe Tricuspid Regurgitation Patients Treated with the Abbott TriClip™ Device (bRIGHT)
Acronym: bRIGHT
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10317
Record Dates: First submitted 2020-07-16; First posted 2020-07-23 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Tricuspid Valve Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Transcatheter heart valve procedure — Transcatheter treatment of TR with Abbott TriClip™.

SUMMARY:
The bRIGHT EU PAS study is an observational real-world study evaluating severe tricuspid regurgitation patients treated with the Abbott TriClip™ device (bRIGHT EU Post-Approval Study).

DETAILED DESCRIPTION:
The TriClip™ bRIGHT EU post-approval study (PAS) study is designed to confirm the safety and performance of the TriClip™ device in a contemporary real-world setting. The bRIGHT PAS study is a prospective, single arm, open-label, multi-center, post market registry, conducted to satisfy condition of CE Marking for the TriClip™.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects (>=18 years age) have severe tricuspid regurgitation and are symptomatic despite medical therapy.
2. Subjects eligible to receive the TriClip™ per the current approved Indications for Use.
3. Subject must provide written informed consent prior to study procedure.

Exclusion Criteria:

1. Subjects participating in another clinical study that may impact the follow-up or results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who have symptomatic severe tricuspid regurgitation despite medical therapy and are eligible to receive the TriClip™ per the current approved Indications For Use.
Sampling Method: Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Acute Procedural Success (APS) | up to 30 days
  The primary endpoint is Acute Procedural Success (APS) defined as successful implantation of the TriClip™ device with resulting TR reduction at least 1 grade at discharge (30-day echocardiogram will be used if discharge is unavailable or uninterpretable). Subjects who die or undergo tricuspid valve surgery before discharge are considered to be an APS failure.

SECONDARY OUTCOMES:
Composite endpoint of all-cause mortality or TR re-intervention | at 1 year follow-up
  The secondary endpoint is a composite endpoint of all-cause mortality or tricuspid valve re-intervention/re-operation at 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Griffin, Study Director — Clinical Program Director
Locations (26):
- Universitätsklinik Graz, Graz, Austria
- Odense University Hospital, Odense, Denmark
- Germany (14):
  - University Hospital Bonn, Bonn, North Rhine-Westphalia
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz, Mainz, Rhineland-Palatinate
  - Leipzig Heart Center, Leipzig, Saxony
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Herz-und Diabetes Zentrum NRW, Bad Oeynhausen
  - Schüchtermann-Schiller´sche Kliniken GmbH & Co. KG, Bad Rothenfelde
  - DRK Kliniken Köpenick, Berlin
  - St.-Johannes-Hospital, Dortmund
  - Elisabeth-Krankenhaus Essen GmbH, Essen
  - Katholisches Marienkrankenhaus GmbH, Hamburg
  - UKE Hamburg (Universitatsklinik Eppendorf), Hamburg
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitätsklinikum Ulm, Ulm
- Italy (3):
  - Maria Cecilia Hospital, Cotignola
  - Azienda Ospedaliera Monaldi, Napoli
  - Universita degli Studi di Padova, Padua
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- Centro Hospitalar Vila Nova de Gaia, Porto, Portugal
- Spain (3):
  - Hospital de Sant Pau, Barcelona, Barcelona
  - Clinical and Provincial Hospital of Barcelona, Barcelona, Barcelona
  - Hospital Álvaro Cunqueiro, Vigo
- Switzerland (2):
  - HerzKlinik Hirslanden - Klinik Hirslanden, Zurich, Canton of Zurich
  - Inselspital Bern, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lurz P, Rommel KP, Schmitz T, Bekeredjian R, Nickenig G, Mollmann H, von Bardeleben RS, Schmeisser A, Atmowihardjo I, Estevez-Loureiro R, Lubos E, Heitkemper M, Peterman K, Lapp H, Donal E. Real-World 1-Year Results of Tricuspid Edge-to-Edge Repair From the bRIGHT Study. J Am Coll Cardiol. 2024 Aug 13;84(7):607-616. doi: 10.1016/j.jacc.2024.05.006. Epub 2024 May 15. PMID 38759905
- [Derived] Lurz P, Besler C, Schmitz T, Bekeredjian R, Nickenig G, Mollmann H, von Bardeleben RS, Schmeisser A, Atmowihardjo I, Estevez-Loureiro R, Lubos E, Heitkemper M, Huang D, Lapp H, Donal E; bRIGHT PAS Principal Investigators. Short-Term Outcomes of Tricuspid Edge-to-Edge Repair in Clinical Practice. J Am Coll Cardiol. 2023 Jul 25;82(4):281-291. doi: 10.1016/j.jacc.2023.05.008. Epub 2023 May 17. PMID 37207923